CLINICAL TRIAL: NCT04866134
Title: A Phase 1b/2, Open-label, Multi-center Study of ERAS-007 (ERK Inhibitor) Administered as Monotherapy or in Combination With ERAS-601 (SHP2 Inhibitor) in Patients With Advanced or Metastatic Solid Tumors (HERKULES-1)
Brief Title: A Study of ERAS-007 as Monotherapy or in Combination With ERAS-601 in Patients With Advanced or Metastatic Solid Tumors
Acronym: HERKULES-1
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Erasca, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERAS-007-01
Record Dates: First submitted 2021-04-24; First posted 2021-04-29 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Advanced or Metastatic Solid Tumors
Keywords: ERK; solid tumor; advanced solid tumor; metastatic solid tumor; neoplasms; solid malignancies; MAPK; SHP2
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Escalation (Part A): ERAS-007 Monotherapy, BID-QW dosing (Experimental): ERAS-007 monotherapy will be administered BID-QW in sequential ascending doses to participants with advanced or metastatic solid tumors until unacceptable toxicity, disease progression, or withdrawal of consent.
  Interventions: Drug: ERAS-007
- Dose Expansion (Part B): ERAS-007 Monotherapy, QW dosing (Experimental): ERAS-007 monotherapy will be administered at 250 mg QW to participants with advanced or metastatic solid tumors that harbor specific molecular alterations.
  Interventions: Drug: ERAS-007
- Dose Expansion (Part C): ERAS-007 Monotherapy, BID-QW dosing (if necessary) (Experimental): Depending on data generated from Part A, ERAS-007 monotherapy may be administered at the BID-QW RD to participants with advanced or metastatic solid tumors that harbor specific molecular alterations.
  Interventions: Drug: ERAS-007
- Dose Escalation (Part D): ERAS-007 BID-QW dosing in combination with ERAS-601 (Experimental): Experimental: Dose Escalation (Part D): ERAS-007 BID-QW dosing in combination with ERAS-601 ERAS-007 will be administered BID-QW in combination with ERAS-601 administered BID 3/1 to study participants with advanced or metastatic solid tumors that harbor specific molecular targets in sequential ascending doses until unacceptable toxicity, disease progression, or withdrawal of consent.
  Interventions: Drug: ERAS-007; Drug: ERAS-601

INTERVENTIONS:
Drug: ERAS-007 — ERAS-007 will be administered orally as specified in Arm description.
Drug: ERAS-601 — ERAS-601 will be administered orally as specified in Arm description.
  Arms: Dose Escalation (Part D): ERAS-007 BID-QW dosing in combination with ERAS-601

SUMMARY:
* To evaluate the safety and tolerability of ERAS-007 monotherapy administered once weekly (QW) and twice daily-once weekly (BID-QW).
* To determine the Maximum Tolerated Dose (MTD) and/or Recommended Dose (RD) of ERAS-007 monotherapy administered BID-QW.
* To characterize the pharmacokinetic (PK) profile of ERAS-007 monotherapy.
* To determine the optimal dose and schedule of ERAS-007 monotherapy.
* To evaluate antitumor activity of ERAS-007 in various solid tumors.
* To evaluate the safety and tolerability of ERAS-007 (BID-QW) and ERAS-601 (twice daily for three weeks on and 1 week off (BID 3/1)) when administered in combination.
* To determine the Maximum Tolerated Dose (MTD) and/or Recommended Dose (RD) of ERAS-007 administered in combination with ERAS-601.
* To characterize the pharmacokinetic (PK) profile of ERAS-007 and ERAS-601 when administered in combination.
* To evaluate antitumor activity of ERAS-007 and ERAS-601 when administered in combination in various solid tumors
* To evaluate antitumor activity of ERAS-007 and ERAS-601 when administered in combination in various solid tumors

DETAILED DESCRIPTION:
This is a Phase 1b/2, open-label, multicenter clinical study of ERAS-007 monotherapy (QW or BID-QW) administered either QW or BID-QWand ERAS-007 (BID-QW) in combination with ERAS-601 (BID 3/1). The monotherapy RD on a weekly schedule has been determined to be 250 mg QW in a previous study. The dose escalation phases of this study will test ERAS-007 monotherapy administered BID-QW as a monotherapy or in combination with ERAS-601 in participants with any solid tumor. The monotherapy RD on a weekly schedule has been determined to be 250 mg QW in a previous study. In parallel, the dose expansion phase of this study will test ERAS-007 monotherapy administered at the RD of 250 mg QW in participants with advanced or metastatic solid tumors harboring specific molecular alterations. Once sufficient safety and PK data are available from the BID-QW dose escalation phase, the Sponsor will then determine the optimal dose and schedule of ERAS-007 administered as a monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Willing and able to give written informed consent.
* Have histologically or cytologically confirmed advanced or metastatic solid tumor with a relevant molecular alteration (as applicable).
* There is no available standard systemic therapy available for the patient's tumor histology and/or molecular biomarker profile; or standard therapy is intolerable, not effective, or not accessible; or patient has refused standard therapy.
* Recovered from all toxicities associated with prior treatment to acceptable baseline status.
* Have ECOG performance status of 0 or 1 with an anticipated life expectancy of > 12 weeks.
* Willing to comply with all protocol-required visits, assessments, and procedures.
* Able to swallow oral medication.

Exclusion Criteria:

* Currently receiving another study therapy or has participated in a study of an investigational agent and received study therapy within 4 weeks of the first dose of ERAS-007.
* Received previous treatment with an ERK inhibitor.
* For participants being considered for ERAS-007 + ERAS-601 (Part D): prior treatment with SHP2 inhibitor.
* For participants being considered for ERAS-007 + ERAS-601 (Part D): documented PTPN11 mutations
* Received prior antineoplastic therapy within < 21 days or 5 half-lives, whichever is shorter.
* Received prior palliative radiation within 7 days of first dose of ERAS 007 or ERAS-601,
* Received previous treatment with a MAPK inhibitor that resulted in discontinuation due to unacceptable toxicity.
* Prior surgery (e.g., gastric bypass surgery, gastrectomy) or gastrointestinal dysfunction (e.g., Crohn's disease, ulcerative colitis, short gut syndrome) that may affect drug absorption.
* Have any underlying medical condition, psychiatric condition, or social situation that, in the opinion of the Investigator, would compromise study administration as per protocol or compromise the assessment of AEs.
* Are pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-05-07 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate safety and tolerability of escalating doses of ERAS-007 BID-QW | Assessed up to 24 months from time of first dose
  Based on adverse events observed
Dose Limiting Toxicities (DLT) | Study Day 1 up to Day 29
  Based on adverse events observed
Maximum tolerated dose (MTD) | Study Day 1 up to Day 29
  Based on adverse events observed
Recommended dose (RD) | Study Day 1 up to Day 29
  Based on adverse events observed
Adverse Events | Assessed up to 24 months from time of first dose
  Incidence and severity of treatment-emergent AEs and serious AEs
Plasma concentration (Cmax) | Study Day 1 up to Day 29
  Maximum plasma concentration of ERAS-007
Time to achieve Cmax (Tmax) | Study Day 1 up to Day 29
  Time to achieve maximum plasma concentration of ERAS-007 and ERAS-601
Area under the curve | Study Day 1 up to Day 29
  Area under the plasma concentration-time curve of ERAS-007 and ERAS-601
Half-life | Study Day 1 up to Day 29
  Half-life of ERAS-007 and ERAS-601

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Assessed up to 24 months from time of first dose
  Based on assessment of radiographic imaging per RECIST version 1.1
Duration of Response (DOR) | Assessed up to 24 months from time of first dose
  Based on assessment of radiographic imaging per RECIST version 1.1
Time to Response (TTR) | Assessed up to 24 months from time of first dose
  Based on assessment of radiographic imaging per RECIST version 1.1

OTHER OUTCOMES:
Pharmacodynamic assessment | Assessed up to 24 months from time of first dose
  Assessment of phosphorylated ERK (pERK) inhibition in isolated PBMCs or tumor tissue by immunoblot, IHC or immunofluorescence.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Lin, M.D., Study Director — Chief Medical Officer
Locations (5):
- United States (5):
  - Sarah Cannon Research Institute (HealthONE), Denver, Colorado
  - Sarah Cannon Research Institute (Florida Cancer Specialists), Sarasota, Florida
  - Sarah Cannon Research Institute (Tennessee Oncology), Nashville, Tennessee
  - Mary Crowley Cancer Research, Dallas, Texas
  - NEXT Oncology, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No